CLINICAL TRIAL: NCT02390895
Title: Prenatal Endoscopic Repair of Fetal Spina Bifida
Acronym: ENDOSPIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P141202; 2014-A01948-39 (Other: ANSM)
Record Dates: First submitted 2015-02-15; First posted 2015-03-18 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Myelomeningocele
Keywords: Minimally-invasive endoscopic repair; fetal surgery; outcome; Foetus
MeSH Terms: conditions — Meningomyelocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Minimally-invasive endoscopic repair (Experimental): endoscopic repair of myelomeningocele before 26 SA
  Interventions: Procedure: endoscopic repair of myelomeningocele before 26 SA

INTERVENTIONS:
Procedure: endoscopic repair of myelomeningocele before 26 SA — prenatal minimally-invasive fetoscopic closure with iii) uterine exteriorization for a minimally-invasive repair under amniotic carbon dioxide insufflation iv) two trocars for the dissection and the cover with one patch or the suture of the skin edges by stitch

SUMMARY:
The purpose of this study is to determine the feasibility of prenatal minimally-invasive fetoscopic closure with i) uterine exteriorization for a minimally-invasive repair under amniotic carbon dioxide insufflation ii) two trocars for the dissection and the cover with one patch or the suture of the skin edges by stitch

DETAILED DESCRIPTION:
Compared with an open approach involving laparotomy and hysterotomy, an endoscopic approach for the prenatal surgery of myelomeningocele offers at least two potential advantages: i) it may reduce the maternal and obstetric morbidity related to the hysterotomy; ii) it may be performed earlier in gestation than open surgery, therefore potentially further reducing exposition of the spinal chord to the intraamniotic environment and thus improving the overall prognosis of the malformation. This study aims to evaluate the feasibility and potential benefits of a minimally invasive endoscopic procedure for the prenatal treatment of myelomeningocele in a single-center trial.

Technically the procedure will be performed through 2 intra-amniotic ports, under fetoscopic visualization and intra-amniotic carbon dioxide insufflation. The defect will be dissected and the cord replaced in the canal. Closure will be performed by suturing paravertebral muscles using a barbed running suture. A Duragen patch will be sutured when primary closure is deemed impossible.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old, with an assumption by health insurance, understanding and speaking French
* A term < or = 26 +0 weeks gestational age
* Single-Pregnancy
* Myelomeningocele with higher-level defect between S1 and T1
* Arnold Chiari anomaly
* No associated anomaly or chromosic anomaly

Exclusion Criteria:

* severe foetal kyphoscoliosis associated
* Increased risk of preterm birth: cervical length <15 mm, history of at least 2 late miscarriages, existing premature rupture of membrane
* placenta previa, accreta or placental abruption
* Maternal obesity with BMI> 35
* Uterine anomalies : large interstitial uterine fibroid, uterine malformation
* maternal infection with a foetal transmission risk: HIV, HBV, HCV
* Maternal contradiction in surgery or anesthesia
* poor social status and/or social isolation
* impossible post-surgery follow-up
* want to have a medical pregnancy termination

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Successful surgery | Before 26 gestational weeks
  Composite criteria:
  1. dissection of the placode
  2. primary coverage or use of a patch
  3. using only endoscopy with two trocars
Neonatal surgery | Day 0 (birth of neonates)
  Need for neonatal surgery
Arnold Chiari anomaly at birth | Day 0 (birth of neonates)
  the existence of an Arnold Chiari anomaly at birth
Ventriculo-peritoneal shunt | Within the 6 months after birth
  Ventriculo-peritoneal shunt within the 6 months after birth
Level of injury | Within the 6 months after birth
Foetal morbidity | From surgery to delivery
  Composite criteria:
  Stillbirth; Premature Rupture of Membranes; Preterm birth; Chorioamnionitis; Hemorrhagic complications during the peri-operative period; Other serious adverse events
Motor lower limb improvement outcomes | Within the 6 months after birth
Maternal morbidity | From surgery to delivery
  Composite criteria:
  Stillbirth; Premature Rupture of Membranes; Preterm birth; Chorioamnionitis; Hemorrhagic complications during the peri-operative period; Other serious adverse events

SECONDARY OUTCOMES:
Neurological development | Within the 12 months after birth
  Composite criteria:
  Motor deficit medullary reflex orthopedic anomalies consequences on perinea and sphincter

CONTACTS AND LOCATIONS:
Overall Officials: Yves Ville, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Julien Stirnemann, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arthuis C, James S, Bussieres L, Hovhannisyan S, Corroenne R, Ville Y, Stirnemann JJ. Laparotomy-Assisted 2-Port Fetoscopic Repair of Spina Bifida Aperta: Report of a Single-Center Experience in Paris, France. Fetal Diagn Ther. 2022;49(9-10):377-384. doi: 10.1159/000525552. Epub 2022 Aug 31. PMID 36044834
- [Background] Kohl T. Percutaneous minimally invasive fetoscopic surgery for spina bifida aperta. Part I: surgical technique and perioperative outcome. Ultrasound Obstet Gynecol. 2014 Nov;44(5):515-24. doi: 10.1002/uog.13430. PMID 24891102
- [Background] Adzick NS, Thom EA, Spong CY, Brock JW 3rd, Burrows PK, Johnson MP, Howell LJ, Farrell JA, Dabrowiak ME, Sutton LN, Gupta N, Tulipan NB, D'Alton ME, Farmer DL; MOMS Investigators. A randomized trial of prenatal versus postnatal repair of myelomeningocele. N Engl J Med. 2011 Mar 17;364(11):993-1004. doi: 10.1056/NEJMoa1014379. Epub 2011 Feb 9. PMID 21306277
- [Background] Degenhardt J, Schurg R, Winarno A, Oehmke F, Khaleeva A, Kawecki A, Enzensberger C, Tinneberg HR, Faas D, Ehrhardt H, Axt-Fliedner R, Kohl T. Percutaneous minimal-access fetoscopic surgery for spina bifida aperta. Part II: maternal management and outcome. Ultrasound Obstet Gynecol. 2014 Nov;44(5):525-31. doi: 10.1002/uog.13389. PMID 24753062
- [Background] Verbeek RJ, Heep A, Maurits NM, Cremer R, Hoving EW, Brouwer OF, van der Hoeven JH, Sival DA. Fetal endoscopic myelomeningocele closure preserves segmental neurological function. Dev Med Child Neurol. 2012 Jan;54(1):15-22. doi: 10.1111/j.1469-8749.2011.04148.x. Epub 2011 Nov 29. PMID 22126123